CLINICAL TRIAL: NCT07225439
Title: Phase I Clinical Trial of Rituximab (Rtx) and Tafasitamab in Combination With Allogeneic NK Cells for Treatment of Relapsed/Refractory (r/r) B-cell Non-Hodgkin Lymphoma
Brief Title: Rituximab (Rtx) + Tafasitamab in Combination With Allogeneic NK Cells for Treatment of Relapsed/Refractory (r/r) B-cell Non-Hodgkin Lymphoma (NHL)
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Paolo Caimi, MD (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor-Investigator, Paolo Caimi, MD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1425
Record Dates: First submitted 2025-11-04; First posted 2025-11-06 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Non Hodgkin Lymphoma; B-cell Non Hodgkin Lymphoma; Diffuse Large B Cell Lymphoma; High-grade B-cell Lymphoma; Primary Mediastinal Large B Cell Lymphoma; Follicular Lymphoma; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Marginal Zone Lymphoma; Mantle Cell Lymphoma
Keywords: NK cells; Natural Killer cells
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell | interventions — Rituximab; resiniferatoxin; tafasitamab; Interleukin-2; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rtx + Tafasitamab in combination with allogeneic NK Cells (Experimental): This arm includes dose escalation for allogeneic NK cells. All other therapies are given according to standard of care. The length of the treatment period is 28 days per cycle. Participants will be expected to complete one cycle and may have the option to complete a second cycle unless there is evidence of disease progression at the end of the first cycle.
  Interventions: Drug: Allogeneic NK cells; Drug: Rituximab; Drug: Tafasitamab; Drug: Interleukin-2; Drug: Fludarabine/cyclophosphamide

INTERVENTIONS:
Drug: Allogeneic NK cells — Allogeneic NK cells are given intravenously (IV) weekly for 3 weeks on Days 0, 7, 14.
  Dose escalation will be conducted using a Bayesian optimal interval (BOIN) design starting at dose level 1 (500 x 106 cells) and proceeding to dose level 2 (1,000 x 106 cells) if criteria are met.
Drug: Rituximab — Rtx is dosed at 375mg/m2 and give once (on Day -5 for Cycle 1 and Day 0 for Cycle 2, if applicable).
  Other Names: Rtx
Drug: Tafasitamab — Tafasitamab is dosed at 12 mg/kg and given intravenously (IV) weekly for 3 weeks on Days 0,7,14).
Drug: Interleukin-2 — Interleukin-2 is dosed at 5 million IU and given weekly for 3 weeks on Days 0,7,14.
Drug: Fludarabine/cyclophosphamide — Fludarabine is dosed at 30 mg/m2/d with dose adjustment for renal function, and cyclophosphamide is dosed at 500 mg/m2/d. These are given on 3 days (Days -5 to -3).
  Other Names: Flu/Cy

SUMMARY:
This research study is for people who have relapsed or refractory B-cell non-Hodgkin's lymphoma (NHL) that has not responded to two or more lines of therapy. The purpose of this study is to identify the recommended dose of allogeneic NK cells in combination with IL-2, Tafasitamab and Rituximab for the treatment of relapsed or refractory B-cell non-Hodgkin's lymphoma.

NK cells are an investigational (experimental) treatment which means they are not approved by the Food and Drug Administration (FDA). NK cells are a type of lymphocyte that's part of the body's natural immune system, and they can kill cancer cells by creating pores in the cancer cell membranes and inducing apoptosis (programmed cell death).

Participants in this study will receive lymphodepleting chemotherapy, as well as Allogeneic NK cells, Tafasitamab and Interleukin-2 (IL-2) by an intravenous (IV) infusion. Participants are expected to complete one cycle, and they may be eligible to complete a second cycle of the same regiment if they have stable disease, partial or complete remission at the end of the first cycle. Participants will be in this study for about 12 months.

DETAILED DESCRIPTION:
More than 80,000 cases of non-Hodgkin lymphoma (NHL) are diagnosed each year in the United States (US), with nearly 20,000 people dying from this group of diseases annually. There are several subgroups of NHL, with the B cell lymphomas being much more common than T-cell lymphomas. B cell lymphomas include multiple different diseases, including some that are more aggressive (like diffuse large B cell lymphoma (DLBCL) and others), as well as those with a slower progression (i.e. indolent lymphomas like follicular lymphoma (FL)). Over the past 20 years, there have been advances in the treatment of most NHL subtypes. However, disease recurrence continues to be frequent and happens in more than a third of people with DLBCL and in most people with indolent lymphomas. A treatment called anti CD19 chimeric antigen receptor T-cell therapies (CAR T-cell) have helped to treat relapsed and primary refractory lymphomas. However, CAR-T cells therapies are limited by the cost and logistics of manufacture. Additionally, relapses are common (40-60%) in people treated with CAR-T cells, and people who experience these relapses have poor survival outcomes.

While CAR-T cells still receive a lot of attention, there is a growing interest in using other strategies including NK cells combined with monoclonal antibodies or molecules developed to activate NK cells against tumors. NK cells are lymphocytes, a type of immune cell, that can naturally fight cancer cells. They are important in fighting cancer and can do so without needing to recognize specific cell markers. Allogeneic, non-HLA-matched NK cells have been found to be safe and not associated with the development of graft-versus-host disease. It is still important to improve the manufacture, application, and efficacy of NK cell therapy. Breakthroughs in ex vivo NK cell expansion have allowed for large doses to be made, which may address some of these limitations.

This study uses a "universal donor" of ex vivo expanded NK cell product that is made at a lab at Case Western Reserve University. These NK cells are "experimental," meaning that they are not approved by the Food and Drug Administration (FDA). Participants in this study will receive these NK cells in addition to other standard cancer treatments for NHL.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosis of B-cell NHL (indolent and aggressive subtypes) including diffuse large B-cell lymphoma not otherwise specified (DLBCL NOS), high grade B-cell lymphoma (HGBCL), primary mediastinal B-cell lymphoma (PMBCL), follicular lymphoma (FL), chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL), marginal zone lymphoma (MZL), and mantle cell lymphoma (MCL)
* Participants must have measurable disease as defined by Lugano 2014 criteria for NHL or iwCLL 2018 criteria for CLL. For NHL, measurable disease is defined as ≥1 measurable lesion (nodal or extra nodal) ≥1.5 cm in longest diameter by CT or PET/CT. For CLL, iwCLL criteria includes: presence of lymphocytosis (e.g., ALC ≥5 × 10⁹/L), lymphadenopathy ≥1.5 cm, and/or disease-related cytopenias (anemia, thrombocytopenia).
* Relapsed and/or refractory after two or more lines of systemic therapy, including prior CD19 and/or CD20 directed therapies
* For participants who have received a prior CD19 or CD20 directed therapy, the presence of CD19 and/or CD20 expression (by flow cytometry and/or immunohistochemistry) must be demonstrated on a post-treatment relapse biopsy
* ECOG Performance Status </= 2
* Preserved organ function as defined by: Total bilirubin </= 1.5X upper limit of normal; AST/ALT </= 2.5 X upper limit of normal; Calculated creatinine clearance >/= 30mL/min estimated by Cockcroft Gualt formula; cardiac ejection fraction >/= 45% and no more than mild/trace pericardial effusion on a recent echocardiogram; and adequate pulmonary function with oxygen saturation >/= 92% on room air.
* Participants must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Second active malignancy (other than non-melanoma skin cancer or carcinoma in situ e.g. cervix, bladder, breast) that would confound interpretation of toxicity assessment or limit survival to prevent evaluation of therapy per discretion of principal investigator. Malignancies treated curatively or with hormonal therapy could be included after discussion with the principal investigator
* Less than 28 days elapsed between prior treatment with investigational agent(s) and study enrollment
* New York Heart Association class III-IV congestive heart failure
* Cardiovascular disorders including unstable angina pectoris, clinically significant cardiac arrhythmias, myocardial infarction or stroke (including transient ischemic attack, or other ischemic event) within 6 months prior to registration
* Known human immunodeficiency virus infection or acquired immunodeficiency syndrome related illness, except well controlled HIV with viral load <200 copies/mL on antiretroviral therapy
* Pregnant or breastfeeding women are excluded from this study because therapy may be associated with the potential for teratogenic or abortifacient effects. Women of childbearing potential must have a negative serum pregnancy test. Because there is an unknown, but potential risk for adverse events in nursing infants' secondary to treatment of the mother with NK cells, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study
* Morphologic and/or cytogenetic features consistent with diagnosis of myelodysplastic syndrome on the most recent bone marrow biopsy prior to initiation of therapy
* Serologic status reflecting active hepatitis B or C infection. Participants that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive participants will be excluded)
* Participants with history of clinically relevant CNS pathology such as epilepsy, seizure disorders, paresis, aphasia, uncontrolled cerebrovascular disease, severe brain injuries, dementia and Parkinson's disease
* Active central nervous system or leptomeningeal involvement by lymphoma. Participants with untreated brain metastases/CNS disease will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurological and other adverse events. Participants with a history of CNS or meningeal involvement must be in a documented remission by CSF evaluation and contrast enhanced MRI imaging for at least 90 days prior to registration
* History of active autoimmune disease (i.e. rheumatoid arthritis, systemic lupus erythematosus) with requirement of systemic immunosuppressive medications other than low dose steroids [i.e. maximum of 15mg prednisone equivalent] within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Up to 42 days
  Non hematologic AEs will be measured during cycle 1 (first 28 days) and hematologic AEs will be measured during the first 42 days for all dose levels. DLTs are graded for severity by the Common Terminology Criteria for Adverse Events v5.0 (CTCAEv5.0) criteria.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 12 months
Timing of adverse events (AEs) | Up to 12 months
Severity of adverse events (AEs) | Up to 12 months
  AE severity will be graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0
Complete response (CR) rate | Day 28
  CR is defined as complete disappearance of all detectable clinical evidence of disease, and disease-related symptoms if present prior to therapy and measured according to the 2014 Lugano Response for Malignant Lymphoma criteria.
Complete response (CR) rate | Day 100
  CR is defined as complete disappearance of all detectable clinical evidence of disease, and disease-related symptoms if present prior to therapy and measured according to the 2014 Lugano Response for Malignant Lymphoma criteria.
Overall response rate (ORR) | Day 28
  ORR is defined as the rate of participants who had CR and partial response (PR). CR is defined as complete disappearance of all detectable clinical evidence of disease, and disease-related symptoms if present prior to therapy and measured according to the 2014 Lugano Response for Malignant Lymphoma criteria. PR is defined as not meeting criteria for CR but having an improvement in symptom criteria specified by the 2014 Lugano Response for Malignant Lymphoma criteria.
Overall response rate (ORR) | Day 100
  ORR is defined as the rate of participants who had CR and partial response (PR). CR is defined as complete disappearance of all detectable clinical evidence of disease, and disease-related symptoms if present prior to therapy and measured according to the 2014 Lugano Response for Malignant Lymphoma criteria. PR is defined as not meeting criteria for CR but having an improvement in symptom criteria specified by the 2014 Lugano Response for Malignant Lymphoma criteria.
Overall survival (OS) | Up to 12 months
  OS is defined as the time from infusion until death from any cause, or until last contact if alive
Event-free survival (EFS) | Up to 12 months
  EFS is defined as the time from infusion until the first occurrence of an event (relapse, progression, or death from any cause), or until last contact if no event occurs.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Caimi, MD, Principal Investigator — Case Comprehensive Cancer Center, Cleveland Clinic
Locations (2):
- United States (2):
  - Case Comprehensive Cancer Center, University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Case Comprehensive Cancer Center, Cleveland Clinic Foundation Taussig Cancer Institute, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Non-Hodgkin Lymphoma - Cancer Stat Facts [Internet]. [cited 2024 Jul 31]. Available from: https://seer.cancer.gov/statfacts/html/nhl.html
- [Background] Coiffier B, Lepage E, Briere J, Herbrecht R, Tilly H, Bouabdallah R, Morel P, Van Den Neste E, Salles G, Gaulard P, Reyes F, Lederlin P, Gisselbrecht C. CHOP chemotherapy plus rituximab compared with CHOP alone in elderly patients with diffuse large-B-cell lymphoma. N Engl J Med. 2002 Jan 24;346(4):235-42. doi: 10.1056/NEJMoa011795. PMID 11807147
- [Background] Duell J, Maddocks KJ, Gonzalez-Barca E, Jurczak W, Liberati AM, De Vos S, Nagy Z, Obr A, Gaidano G, Abrisqueta P, Kalakonda N, Andre M, Dreyling M, Menne T, Tournilhac O, Augustin M, Rosenwald A, Dirnberger-Hertweck M, Weirather J, Ambarkhane S, Salles G. Long-term outcomes from the Phase II L-MIND study of tafasitamab (MOR208) plus lenalidomide in patients with relapsed or refractory diffuse large B-cell lymphoma. Haematologica. 2021 Sep 1;106(9):2417-2426. doi: 10.3324/haematol.2020.275958. PMID 34196165
- [Background] Sehn LH, Herrera AF, Flowers CR, Kamdar MK, McMillan A, Hertzberg M, Assouline S, Kim TM, Kim WS, Ozcan M, Hirata J, Penuel E, Paulson JN, Cheng J, Ku G, Matasar MJ. Polatuzumab Vedotin in Relapsed or Refractory Diffuse Large B-Cell Lymphoma. J Clin Oncol. 2020 Jan 10;38(2):155-165. doi: 10.1200/JCO.19.00172. Epub 2019 Nov 6. PMID 31693429
- [Background] Caimi PF, Ai W, Alderuccio JP, Ardeshna KM, Hamadani M, Hess B, Kahl BS, Radford J, Solh M, Stathis A, Zinzani PL, Havenith K, Feingold J, He S, Qin Y, Ungar D, Zhang X, Carlo-Stella C. Loncastuximab tesirine in relapsed or refractory diffuse large B-cell lymphoma (LOTIS-2): a multicentre, open-label, single-arm, phase 2 trial. Lancet Oncol. 2021 Jun;22(6):790-800. doi: 10.1016/S1470-2045(21)00139-X. Epub 2021 May 11. PMID 33989558
- [Background] Byrd JC, Harrington B, O'Brien S, Jones JA, Schuh A, Devereux S, Chaves J, Wierda WG, Awan FT, Brown JR, Hillmen P, Stephens DM, Ghia P, Barrientos JC, Pagel JM, Woyach J, Johnson D, Huang J, Wang X, Kaptein A, Lannutti BJ, Covey T, Fardis M, McGreivy J, Hamdy A, Rothbaum W, Izumi R, Diacovo TG, Johnson AJ, Furman RR. Acalabrutinib (ACP-196) in Relapsed Chronic Lymphocytic Leukemia. N Engl J Med. 2016 Jan 28;374(4):323-32. doi: 10.1056/NEJMoa1509981. Epub 2015 Dec 7. PMID 26641137
- [Background] Eichhorst B, Niemann CU, Kater AP, Furstenau M, von Tresckow J, Zhang C, Robrecht S, Gregor M, Juliusson G, Thornton P, Staber PB, Tadmor T, Lindstrom V, da Cunha-Bang C, Schneider C, Poulsen CB, Illmer T, Schottker B, Nosslinger T, Janssens A, Christiansen I, Baumann M, Frederiksen H, van der Klift M, Jager U, Leys MBL, Hoogendoorn M, Lotfi K, Hebart H, Gaska T, Koene H, Enggaard L, Goede J, Regelink JC, Widmer A, Simon F, De Silva N, Fink AM, Bahlo J, Fischer K, Wendtner CM, Kreuzer KA, Ritgen M, Bruggemann M, Tausch E, Levin MD, van Oers M, Geisler C, Stilgenbauer S, Hallek M; GCLLSG, the HOVON and Nordic CLL Study Groups, the SAKK, the Israeli CLL Association, and Cancer Trials Ireland. First-Line Venetoclax Combinations in Chronic Lymphocytic Leukemia. N Engl J Med. 2023 May 11;388(19):1739-1754. doi: 10.1056/NEJMoa2213093. PMID 37163621
- [Background] ASCO Daily News [Internet]. [cited 2024 Jul 31]. How Do CAR T Cells Fit Into the Evolving Non-Hodgkin Lymphoma Treatment Landscape? Available from: https://dailynews.ascopubs.org/doi/10.1200/ADN.24.201682
- [Background] Di Blasi R, Le Gouill S, Bachy E, Cartron G, Beauvais D, Le Bras F, Gros FX, Choquet S, Bories P, Feugier P, Casasnovas O, Bay JO, Mohty M, Joris M, Gastinne T, Sesques P, Tudesq JJ, Vercellino L, Morschhauser F, Gat E, Broussais F, Houot R, Thieblemont C. Outcomes of patients with aggressive B-cell lymphoma after failure of anti-CD19 CAR T-cell therapy: a DESCAR-T analysis. Blood. 2022 Dec 15;140(24):2584-2593. doi: 10.1182/blood.2022016945. PMID 36122385
- [Background] Gu T, Zhu M, Huang H, Hu Y. Relapse after CAR-T cell therapy in B-cell malignancies: challenges and future approaches. J Zhejiang Univ Sci B. 2022 Oct 15;23(10):793-811. doi: 10.1631/jzus.B2200256. PMID 36226535
- [Background] Derigs P, Bethge WA, Kramer I, Holtick U, von Tresckow B, Ayuk F, Penack O, Vucinic V, von Bonin M, Baldus C, Mougiakakos D, Wulf G, Schnetzke U, Stelljes M, Fante M, Schroers R, Kroeger N, Dreger P; German Lymphoma Alliance and the German Registry for Stem Cell Transplantation. Long-Term Survivors after Failure of Chimeric Antigen Receptor T Cell Therapy for Large B Cell Lymphoma: A Role for Allogeneic Hematopoietic Cell Transplantation? A German Lymphoma Alliance and German Registry for Stem Cell Transplantation Analysis. Transplant Cell Ther. 2023 Dec;29(12):750-756. doi: 10.1016/j.jtct.2023.09.008. Epub 2023 Sep 13. PMID 37709204
- [Background] Grossenbacher SK, Aguilar EG, Murphy WJ. Leveraging natural killer cells for cancer immunotherapy. Immunotherapy. 2017 May;9(6):487-497. doi: 10.2217/imt-2017-0013. PMID 28472904
- [Background] Olson JA, Leveson-Gower DB, Gill S, Baker J, Beilhack A, Negrin RS. NK cells mediate reduction of GVHD by inhibiting activated, alloreactive T cells while retaining GVT effects. Blood. 2010 May 27;115(21):4293-301. doi: 10.1182/blood-2009-05-222190. Epub 2010 Mar 16. PMID 20233969